CLINICAL TRIAL: NCT03558061
Title: A Single Arm Open-Label Study to Evaluate the Therapeutic Effects and Safety of a 6-Week Treatment Regimen of ALK4290 in Patients With Newly Diagnosed Wet Age-Related Macular Degeneration (wAMD)
Brief Title: Evaluate the Effects and Safety of ALK4290 in Patients With Newly Diagnosed Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK4290-201
Record Dates: First submitted 2018-05-15; First posted 2018-06-15 (Actual); Results first posted 2020-08-28 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2018-12

CONDITIONS: Wet Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active (Experimental): ALK4290 800 mg daily
  Interventions: Drug: ALK4290

INTERVENTIONS:
Drug: ALK4290 — ALK4290 400 mg tablet twice a day
  Other Names: AKST4290; BI 144807

SUMMARY:
This study will evaluate the therapeutic effects and safety of 800 mg ALK4290 administered daily over a 6-week dosing period in newly diagnosed patients with wet age-related macular degeneration (wAMD).

DETAILED DESCRIPTION:
This study is designed to evaluate the therapeutic effects and safety of oral ALK4290 administered at 800 mg daily over a 6-week dosing period in newly diagnosed (treatment naïve) patients with wAMD. The study agent will be orally self-administered. All subjects will receive the study agent, ALK4290. This study does not contain a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with newly diagnosed active CNV secondary to AMD, diagnosed by a retinal specialist with all the following characteristics and ophthalmic inclusion criteria applied to the study eye:

  * No prior treatment for wAMD in the study eye and no current or planned concomitant intravitreal anti-VEGF treatment in the fellow eye
  * Central subfield retinal thickness ≥ 250 microns on SD-OCT (exclusive of subretinal pigment epithelial fluid, inclusive of SRF)
  * Presence of SRF and/or IRF on SD-OCT
  * Any active CNV with subfoveal leakage as determined by FA
  * Total lesion size not greater than 12 disc areas on FA
  * If present, subretinal hemorrhage must comprise < 50% of the total lesion area on FA
  * No subfoveal fibrosis or atrophy on FA
* BCVA letter score, as measured by ETDRS in the study eye, between 70 and 24 letters, inclusive, at screening
* Patients 50 years of age or older at screening visit 1
* Body mass index (BMI) between18 and ≤ 40 at screening visit 1
* Female subjects must not be pregnant or breastfeeding. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry.
* Signed informed consent consistent with ICH-GCP guidelines and local legislation prior to participation in the trial, which includes medication washout and restrictions

Exclusion Criteria:

* Previous participation in any studies of investigational drugs within 1 month preceding screening visit
* Any form of macular degeneration that is not age-related (e.g., Best's disease, Stargardt's disease, Sorsby's disease, etc.)
* Additional eye disease in the study eye that could compromise BCVA (i.e., uncontrolled glaucoma (intraocular pressure > 24) with visual field loss, clinically significant diabetic maculopathy, history of ischemic optic neuropathy or retinal vascular occlusion, vitreomacular traction, monocular vision, or genetic disorders such as retinitis pigmentosa; high myopia > 8 diopters)
* The presence of polypoidal choroidal vasculopathy (PCV) or retinal angiomatous proliferation (RAP) in the study eye
* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with fundus photography/FA or SD-OCT
* Intraocular surgery in the study eye within 3 months prior to screening
* Aphakia or total absence of the posterior capsule (yttrium aluminum garnet (YAG) laser capsulotomy permitted, a minimum of 1 month prior to enrollment) in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2018-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (5):
- Hungary (5):
  - Jahn Ferenc South-Pest Hospital and Clinic, Budapest
  - Borsod-Abauj-Zemplen County Hospital and Teaching Hospital, Miskolc
  - Szabolcs-Szatmar-Bereg County Hospital and University Hospital, Nyíregyháza
  - University of Szeged Faculty of Medicine, Szeged
  - Markusovszky University Teaching Hospital, Szombathely

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 8
  Poland | 22

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity (BCVA)
Description: Mean change in BCVA letter score as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) method. The ETDRS chart assesses changes in vision based on the number of letters correctly read by the subject.
Time Frame: Baseline to 6 weeks
Population: Evaluable Set
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Active
Number analyzed (Participants) | 29
letters | 7.0 (12.51)

2. Secondary Outcome: Incidence of Treatment-emergent Adverse Events (Safety)
Description: Treatment-emergent adverse events identified by the Common Terminology Criteria for Adverse Events (CTCAE v4.03)
Time Frame: Baseline to 10 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 30
Participants | 14

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 14/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=30)
Visual acuity reduced (Eye disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Cystitis (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03558061/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT03558061/SAP_001.pdf